CLINICAL TRIAL: NCT03762616
Title: Urology San Antonio MRI/MicroUS Comparison
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Exact Imaging (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: EVU-2018-001
Record Dates: First submitted 2018-11-27; First posted 2018-12-04 (Actual); Results first posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer
Keywords: multiparametric MRI; micro-ultrasound; prostate biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigator performing the micro-ultrasound biopsy will be blinded to the MRI report, and the investigator performing the MRI targeted biopsy will be blinded to the micro-ultrasound images and targets.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Micro-Ultrasound Biopsy (Experimental)
  Interventions: Diagnostic Test: Micro-ultrasound targeted biopsy
- MRI Targeted Biopsy (Experimental)
  Interventions: Diagnostic Test: mpMRI targeted biopsy

INTERVENTIONS:
Diagnostic Test: Micro-ultrasound targeted biopsy — Micro-ultrasound targeted biopsy using the ExactVu micro-ultrasound system
  Arms: Micro-Ultrasound Biopsy
Diagnostic Test: mpMRI targeted biopsy — Multiparametric MRI targeted biopsy using software assisted MRI/US fusion
  Arms: MRI Targeted Biopsy

SUMMARY:
This study compares micro-ultrasound image targeted prostate biopsy with multi-parametric MRI targeted biopsy in men indicated for prostate biopsy due to suspicion of prostate cancer. Both imaging techniques will be applied to each subject and compared, along with systematic biopsy.

DETAILED DESCRIPTION:
The investigational protocol describes a study designed to compare ultra-high resolution transrectal micro-ultrasound (micro-US), and multi-parametric MRI (mpMRI). These modalities are both used clinically to identify targets for prostate biopsy, however little data is available to compare their sensitivity. While mpMRI is used clinically to identify targets for biopsy, it is not used for real-time biopsy guidance due to challenges performing the biopsy procedure within the MRI gantry. Instead, targets identified on mpMRI are sampled during transrectal ultrasound guided biopsy as part of the prostate biopsy procedure, often using software assisted fusion products. For this investigation, the biopsy procedure will be guided by transrectal micro-US (current standard of care at Urology San Antonio), and will include systematic (standard, random, extended sextant) plus image-guided prostate biopsies among men with clinical suspicion of prostate cancer and an indication for prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Men presenting for prostate biopsy due to clinical suspicion of prostate cancer
2. 40-75 years old
3. Available mpMRI images and report, performed according to the PI-RADS v2 standard

Exclusion Criteria:

1. Men with anorectal abnormalities preventing TRUS-guided prostate biopsy
2. Men who are unable to provide their own informed consent
3. Prostate volume on MRI > 100cc

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Talley, MD, Principal Investigator — Urology San Antonio
Locations (1):
- Urology San Antonio - Pasteur Plaza Surgery Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Micro-ultrasound Biopsy Then MRI Biopsy: Micro-ultrasound targeted biopsy: Micro-ultrasound targeted biopsy using the ExactVu micro-ultrasound system Followed in the same session by MRI biopsy by a second blinded operator
Period: Overall Study
Arm/Group | Micro-ultrasound Biopsy Then MRI Biopsy
Started | 120
Completed | 118
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Groups:
- Micro-ultrasound Biopsy Then MRI Biopsy: Micro-ultrasound targeted biopsy: Micro-ultrasound targeted biopsy using the ExactVu micro-ultrasound system Followed in the same session by... mpMRI targeted biopsy: Multiparametric MRI targeted biopsy using software assisted MRI/US fusion
Arm/Group | Micro-ultrasound Biopsy Then MRI Biopsy
Number analyzed (Participants) | 118
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67 [62 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 118
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 118

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Cancer
Description: Comparison of subject-level detection rate of clinically significant cancer (csPCa, defined as Grade Group 2 or higher) between micro-ultrasound targeted biopsy and mpMRI targeted biopsy.
Time Frame: At time of biopsy
Measure: Count of Participants; unit: Participants
Groups:
- Micro-ultrasound Biopsy: Micro-ultrasound biopsy: Micro-ultrasound biopsy using the ExactVu micro-ultrasound system
Arm/Group | Micro-ultrasound Biopsy | MRI Targeted Biopsy
Number analyzed (Participants) | 118 | 118
Participants | 38 | 31

ADVERSE EVENTS:
Time Frame: During biopsy procedure
Arm/Group | Micro-ultrasound Targeted Biopsy | MRI Targeted Biopsy
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/118
Serious Adverse Events (participants affected / at risk) | 0/118 | 0/118
Other Adverse Events (participants affected / at risk) | 0/118 | 0/118

LIMITATIONS AND CAVEATS:
Due to issues with marking of targeted samples the primary endpoint was modified to distinguish between the two devices used in the arms rather than biopsy annotations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT03762616/Prot_SAP_000.pdf